CLINICAL TRIAL: NCT01892228
Title: Pilot Study of Immediate HIV Treatment by Means of "One-stop Service" in Hospital in Guangxi, China
Brief Title: Pilot Study of Immediate HIV Treatment in Guangxi, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Treat-All HIV Pilot
Record Dates: First submitted 2013-05-18; First posted 2013-07-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2013-06

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome
Keywords: antiretroviral therapy; education; mortality
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Two counties: Zhongshan and Pubei (Experimental): Immediate post-screening treatment education for HIV-positive participants residing in the Zhongshan and Pubei pilot sites in the "Treat-All" HIV Pilot Program
  Interventions: Behavioral: Immediate post-screening treatment education

INTERVENTIONS:
Behavioral: Immediate post-screening treatment education — immediate treatment education after screening to decrease time from initial HIV screening to treatment implementation

SUMMARY:
The aim of the study is to measure the effectiveness of a pilot program in Guangxi, China to decrease mortality related to HIV.

The study's proposed mechanism of decreasing mortality rates is to shorten the time between initial HIV screening and ART implementation to within two weeks.

The study population consists of participants who received an initial HIV infection diagnosis within the study period. Medical institutions will provide "one-stop services" by following detailed guidelines regarding reporting of positive HIV antibody screenings, further testing procedures, and treatment referrals in accordance with a pre-determined timetable. In addition, additional strategies focusing on policy development, medical personnel training, and a broad general public education campaign will be implemented.

Main assessment measures are HIV-related mortality rates, treatment coverage, or other health outcomes.

DETAILED DESCRIPTION:
The aim of the study is to measure the effectiveness of a pilot program in Guangxi, China to decrease mortality related to HIV/AIDS. In past years, Guangxi has experienced a relatively high rate of late HIV diagnoses, which has contributed to a significant proportion of HIV-related deaths occurring in the same year of initial diagnosis. The study's proposed mechanism of decreasing mortality rates is to shorten the time between initial HIV screening and ART implementation to within two weeks.

Two pilot sites were selected based on past core assessment indicators. The study population consists of participants who received an initial HIV infection diagnosis within the study period. Medical institutions will provide "one-stop services" by following detailed guidelines regarding reporting of positive HIV antibody screenings, further testing procedures, and treatment referrals in accordance with a pre-determined timetable. In addition, additional strategies focusing on policy development, medical personnel training, and a broad general public education campaign will be implemented.

The study will be performed from July,2012 to July,2015. Main assessment measures are HIV-related mortality rates, treatment coverage, or other health outcomes.

1. HIV-related mortality rates of participants who are newly diagnosed during the study period Numerator: Number of all-cause deaths during the study period Denominator: Number of HIV infected patients followed during the study period.
2. Percentage of newly diagnosed HIV-infected participants who receive ART Numerator: Number of patients who are diagnosed with HIV and initiate ART during the study period Denominator: Number of newly reported HIV cases during the study period

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of HIV infection as defined by having positive HIV antibody screening results between July 1, 2012 and July 1, 2015 OR
* Having a current residential address inside of pilot site limits

Exclusion criteria:

* Current residing outside of the borders of the designated study sites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
mortality | 12 months
  HIV-related mortality rates of participants who are newly diagnosed during the study period Numerator: Number of all-cause deaths during the study period Denominator: Number of HIV infected patients followed during the study period.
ART treatment coverage | 12 months
  Percentage of newly diagnosed HIV-infected participants who receive ART Numerator: Number of patients who are diagnosed with HIV and initiate ART during the study period Denominator: Number of newly reported HIV cases during the study period

SECONDARY OUTCOMES:
mortality | 36 months
  mortality rates of participants who are newly diagnosed during the study period Numerator: Number of all-cause deaths during the study period Denominator: Number of HIV infected patients followed during the study period.
ART treatment coverage | 36 months
  Percentage of newly diagnosed HIV-infected participants who receive ART Numerator: Number of patients who are diagnosed with HIV and initiate ART during the study period Denominator: Number of newly reported HIV cases during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, PhD, Study Chair — National Center for AIDS/STD Control and Prevention
Locations (2):
- China (2):
  - Pubei Center for Disease Control, Xiaojiang, Guangxi
  - Zhongshan Center for Disease Control, Zhongshan